CLINICAL TRIAL: NCT00704379
Title: Treatment Strategy to Prevent Mood Disorders Following Traumatic Brain Injury
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Ricardo Jorge, MD, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R01NS055827 (NIH); 1R01NS055827-01A2 (NIH)
Record Dates: First submitted 2008-06-20; First posted 2008-06-24 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury; TBI; mood disorders; anxiety disorders; community reintegration; executive function; sertraline; diffusion tensor imaging
MeSH Terms: conditions — Brain Injuries, Traumatic; Mood Disorders; Anxiety Disorders | interventions — Sertraline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo will be given in a double blind fashion via an equal number of tablets (identical to the sertraline tablets) administered once daily.
  Interventions: Drug: Placebo
- Sertraline (Experimental): Sertraline will be given in a double blind fashion via tablets administered once daily. Once stabilized in the targeted dosage (100 mg per day), sertraline serum levels will be monitored twice during the course of the intervention.
  Interventions: Drug: Sertraline

INTERVENTIONS:
Drug: Placebo — an inactive substance
  Arms: Placebo
Drug: Sertraline — Sertraline and placebo will be given in a double blind fashion via an equal number of identical tablets administered once daily. Once stabilized in the targeted dosage (100 mg per day), sertraline serum levels will be monitored twice during the course of the intervention. Blood samples will be obtained randomly, one during the first and one during the second trimesters of the protocol.
  Other Names: Zoloft
  Arms: Sertraline

SUMMARY:
The purpose of this study is to examine the efficacy of sertraline to prevent the onset of mood and anxiety disorders during the first six months after traumatic brain injury.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is a leading cause of death and disability among young adults. Mood disorders are the most frequent psychiatric complication of TBI, and have a large impact on family functioning, interpersonal relationships, and ability to return to work or school. Furthermore, a significant proportion of these disorders will progress to more chronic and treatment refractory forms. In spite of their clinical relevance, mood and anxiety disorders remain largely unrecognized and not adequately treated, contributing to greater disability and decreased participation in the aftermath of TBI.

The goals of this study are to learn more about how people recover from brain injury and to evaluate the effect of sertraline (also known as Zoloft) compared to placebo (an inactive substance) in preventing the occurrence of emotional and behavioral problems-such as depression, lack of motivation, anxiety, irritability or aggressive outbursts-following TBI.

In the study, a group of 104 participants with TBI-recruited immediately after resolution of posttraumatic amnesia-will be randomly assigned to receive six months of double-blind treatment with sertraline or placebo.

This study will determine how these emotional and behavioral problems influence thinking, physical recovery, and return to a productive life six months after brain injury. Researchers will also determine if certain brain changes can predict the occurrence of behavioral problems and if treatment with sertraline can prevent them. Additionally, the researchers will examine the effect of sertraline on frequent post-TBI behavioral disorders such as aggression, impulsivity, poor decision making and apathetic symptoms.

Magnetic resonance imaging (MRI)-based volumetry and diffusion tensor imaging will be used to examine the structural correlates of mood and anxiety disorders and to evaluate them as biological predictors of treatment response and community reintegration. The researchers hypothesize that early preventive treatment with sertraline will reduce mood and behavioral symptoms, prevent the occurrence of structural and functional brain changes associated with the onset of mood disorders, increase access to and participation in rehabilitation programs for TBI, and, consequently, improve psychosocial outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or over.
* Meeting the Center for Disease Control (CDC) criteria for TBI.
* Mild, Moderate, or Severe TBI as categorized by initial Glasgow Coma Scale (GCS) scores 13 to 15, 9 to 12, or 3 to 8, respectively.
* Complete recovery from Post Traumatic Amnesia (PTA) within 4 weeks of the traumatic episode.

Exclusion Criteria:

* Penetrating head injuries.
* Clinical or neuro-radiological evidence of associate spinal cord injury.
* Patients with severe comprehension deficits (i.e., those who are not able to complete part II of the Token Test) that precludes a thorough neuropsychiatric evaluation.
* Presence of Diagnostic and Statistical Manual IV defined mood, anxiety or psychotic disorder at the time of enrollment to the study. However, patients with a history of alcohol abuse or alcohol dependence during the year preceding TBI will be included in the study.
* Patients who were taking antidepressants at the time of TBI or during a six month period prior to the traumatic event.
* Patients who have failed an adequate previous trial with sertraline or had side effects that prompted the discontinuation of this medication.
* Pregnant women or women that plan to become pregnant during the period of the study.
* Severe complicating illness such as neoplastic disease or uncompensated heart, renal or liver failure.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2008-06; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo E. Jorge, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Background] Arciniegas DB, Topkoff J, Silver JM. Neuropsychiatric Aspects of Traumatic Brain Injury. Curr Treat Options Neurol. 2000 Mar;2(2):169-186. doi: 10.1007/s11940-000-0017-y. PMID 11096746
- [Background] Fann JR, Burington B, Leonetti A, Jaffe K, Katon WJ, Thompson RS. Psychiatric illness following traumatic brain injury in an adult health maintenance organization population. Arch Gen Psychiatry. 2004 Jan;61(1):53-61. doi: 10.1001/archpsyc.61.1.53. PMID 14706944
- [Background] Silver JM, Hales RE, Yudofsky SC. Psychopharmacology of depression in neurologic disorders. J Clin Psychiatry. 1990 Jan;51 Suppl:33-9. PMID 2404002
- [Background] Jorge RE, Robinson RG, Moser D, Tateno A, Crespo-Facorro B, Arndt S. Major depression following traumatic brain injury. Arch Gen Psychiatry. 2004 Jan;61(1):42-50. doi: 10.1001/archpsyc.61.1.42. PMID 14706943
- [Background] Fann JR, Uomoto JM, Katon WJ. Sertraline in the treatment of major depression following mild traumatic brain injury. J Neuropsychiatry Clin Neurosci. 2000 Spring;12(2):226-32. doi: 10.1176/jnp.12.2.226. PMID 11001601
- [Background] Graham DI, McIntosh TK, Maxwell WL, Nicoll JA. Recent advances in neurotrauma. J Neuropathol Exp Neurol. 2000 Aug;59(8):641-51. doi: 10.1093/jnen/59.8.641. PMID 10952055
- [Background] McIntosh TK, Saatman KE, Raghupathi R, Graham DI, Smith DH, Lee VM, Trojanowski JQ. The Dorothy Russell Memorial Lecture. The molecular and cellular sequelae of experimental traumatic brain injury: pathogenetic mechanisms. Neuropathol Appl Neurobiol. 1998 Aug;24(4):251-67. doi: 10.1046/j.1365-2990.1998.00121.x. PMID 9775390
- [Background] Buki A, Povlishock JT. All roads lead to disconnection?--Traumatic axonal injury revisited. Acta Neurochir (Wien). 2006 Feb;148(2):181-93; discussion 193-4. doi: 10.1007/s00701-005-0674-4. Epub 2005 Dec 20. PMID 16362181
- [Background] Manji HK, Quiroz JA, Sporn J, Payne JL, Denicoff K, A Gray N, Zarate CA Jr, Charney DS. Enhancing neuronal plasticity and cellular resilience to develop novel, improved therapeutics for difficult-to-treat depression. Biol Psychiatry. 2003 Apr 15;53(8):707-42. doi: 10.1016/s0006-3223(03)00117-3. PMID 12706957
- [Background] Warner-Schmidt JL, Duman RS. Hippocampal neurogenesis: opposing effects of stress and antidepressant treatment. Hippocampus. 2006;16(3):239-49. doi: 10.1002/hipo.20156. PMID 16425236
- [Background] Duman RS, Monteggia LM. A neurotrophic model for stress-related mood disorders. Biol Psychiatry. 2006 Jun 15;59(12):1116-27. doi: 10.1016/j.biopsych.2006.02.013. Epub 2006 Apr 21. PMID 16631126
- [Background] Santarelli L, Saxe M, Gross C, Surget A, Battaglia F, Dulawa S, Weisstaub N, Lee J, Duman R, Arancio O, Belzung C, Hen R. Requirement of hippocampal neurogenesis for the behavioral effects of antidepressants. Science. 2003 Aug 8;301(5634):805-9. doi: 10.1126/science.1083328. PMID 12907793
- [Background] Normann C, Schmitz D, Furmaier A, Doing C, Bach M. Long-term plasticity of visually evoked potentials in humans is altered in major depression. Biol Psychiatry. 2007 Sep 1;62(5):373-80. doi: 10.1016/j.biopsych.2006.10.006. Epub 2007 Jan 19. PMID 17240361
- [Background] Sheline YI, Barch DM, Donnelly JM, Ollinger JM, Snyder AZ, Mintun MA. Increased amygdala response to masked emotional faces in depressed subjects resolves with antidepressant treatment: an fMRI study. Biol Psychiatry. 2001 Nov 1;50(9):651-8. doi: 10.1016/s0006-3223(01)01263-x. PMID 11704071
- [Background] Anand A, Li Y, Wang Y, Wu J, Gao S, Bukhari L, Mathews VP, Kalnin A, Lowe MJ. Antidepressant effect on connectivity of the mood-regulating circuit: an FMRI study. Neuropsychopharmacology. 2005 Jul;30(7):1334-44. doi: 10.1038/sj.npp.1300725. PMID 15856081
- [Background] Bechara A, Damasio H, Tranel D, Damasio AR. The Iowa Gambling Task and the somatic marker hypothesis: some questions and answers. Trends Cogn Sci. 2005 Apr;9(4):159-62; discussion 162-4. doi: 10.1016/j.tics.2005.02.002. PMID 15808493
- [Background] Huisman TA, Schwamm LH, Schaefer PW, Koroshetz WJ, Shetty-Alva N, Ozsunar Y, Wu O, Sorensen AG. Diffusion tensor imaging as potential biomarker of white matter injury in diffuse axonal injury. AJNR Am J Neuroradiol. 2004 Mar;25(3):370-6. PMID 15037457
- [Background] Salmond CH, Menon DK, Chatfield DA, Williams GB, Pena A, Sahakian BJ, Pickard JD. Diffusion tensor imaging in chronic head injury survivors: correlations with learning and memory indices. Neuroimage. 2006 Jan 1;29(1):117-24. doi: 10.1016/j.neuroimage.2005.07.012. Epub 2005 Aug 9. PMID 16084738
- [Background] Le TH, Mukherjee P, Henry RG, Berman JI, Ware M, Manley GT. Diffusion tensor imaging with three-dimensional fiber tractography of traumatic axonal shearing injury: an imaging correlate for the posterior callosal
- [Background] Jorge R, Robinson RG. Mood disorders following traumatic brain injury. NeuroRehabilitation. 2002;17(4):311-24. No abstract available. PMID 12547979
- [Background] Jorge RE, Robinson RG, Arndt S. Are there symptoms that are specific for depressed mood in patients with traumatic brain injury? J Nerv Ment Dis. 1993 Feb;181(2):91-9. doi: 10.1097/00005053-199302000-00004. PMID 8426177
- [Background] Jorge RE, Robinson RG, Arndt SV, Forrester AW, Geisler F, Starkstein SE. Comparison between acute- and delayed-onset depression following traumatic brain injury. J Neuropsychiatry Clin Neurosci. 1993 Winter;5(1):43-9. doi: 10.1176/jnp.5.1.43. PMID 8428134
- [Background] Jorge RE, Robinson RG, Arndt SV, Starkstein SE, Forrester AW, Geisler F. Depression following traumatic brain injury: a 1 year longitudinal study. J Affect Disord. 1993 Apr;27(4):233-43. doi: 10.1016/0165-0327(93)90047-n. PMID 8509524
- [Background] Jorge RE, Robinson RG, Starkstein SE, Arndt SV. Depression and anxiety following traumatic brain injury. J Neuropsychiatry Clin Neurosci. 1993 Fall;5(4):369-74. doi: 10.1176/jnp.5.4.369. PMID 8286933
- [Background] Jorge RE, Robinson RG, Starkstein SE, Arndt SV. Influence of major depression on 1-year outcome in patients with traumatic brain injury. J Neurosurg. 1994 Nov;81(5):726-33. doi: 10.3171/jns.1994.81.5.0726. PMID 7931619
- [Background] Jorge RE, Robinson RG, Starkstein SE, Arndt SV, Forrester AW, Geisler FH. Secondary mania following traumatic brain injury. Am J Psychiatry. 1993 Jun;150(6):916-21. doi: 10.1176/ajp.150.6.916. PMID 8494069
- [Background] Jorge R, Robinson RG. Mood disorders following traumatic brain injury. Int Rev Psychiatry. 2003 Nov;15(4):317-27. doi: 10.1080/09540260310001606700. PMID 15276953
- [Background] Jorge RE, Starkstein SE. Pathophysiologic aspects of major depression following traumatic brain injury. J Head Trauma Rehabil. 2005 Nov-Dec;20(6):475-87. doi: 10.1097/00001199-200511000-00001. PMID 16304485
- [Background] Tateno A, Jorge RE, Robinson RG. Pathological laughing and crying following traumatic brain injury. J Neuropsychiatry Clin Neurosci. 2004 Fall;16(4):426-34. doi: 10.1176/jnp.16.4.426. PMID 15616168
- [Derived] Jorge RE, Acion L, Burin DI, Robinson RG. Sertraline for Preventing Mood Disorders Following Traumatic Brain Injury: A Randomized Clinical Trial. JAMA Psychiatry. 2016 Oct 1;73(10):1041-1047. doi: 10.1001/jamapsychiatry.2016.2189. PMID 27626622

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo (i.e., an inactive substance) was given in a double blind fashion via an equal number of tablets (identical to the sertraline tablets) administered once daily.
- Sertraline: Sertraline (other name: Zoloft) was administered in a double blind fashion via tablets administered once daily. Targeted dosage: 100 mg/day.
Period: Overall Study
Arm/Group | Placebo | Sertraline
Started | 46 | 48
Completed | 39 | 41
Not Completed | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Sertraline | Total
Number analyzed (Participants) | 46 | 48 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.91 (18.24) | 49.98 (20.05) | 52.39 (19.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 22 | 38
  Male | 30 | 26 | 56

OUTCOME MEASURES:

1. Primary Outcome: Time to Onset of Diagnostic and Statistical Manual (DSM) IV Defined Mood and Anxiety Disorders Associated With Traumatic Brain Injury (TBI)
Description: Following the DSM-IV (now updated by the DSM-5), depressive disorders associated with TBI are categorized as Mood Disorder Due to Another Medical Condition with subtypes: 1) With major depressive-like episode (if the full criteria for a major depressive episode [MDE] are met) or 2) With depressive features (prominent depressed mood but full criteria for a MDE are not met); and 3) with mixed features (e.g. significant irritability, pressured speech and formal thought disorder).
  On the other hand, bipolar and related disorders due to TBI are subdivided in: 1) with manic or hypomanic like episode; 2) with manic features; and 3) with mixed features.
  A similar conceptual framework has been used to define Anxiety Disorder due to another Medical Condition, in this case, TBI. According to DSM-IV/DSM-5, such diagnosis can be made when, besides an evident pathophysiological relationship with TBI, panic attacks or generalized anxiety are the prominent features of the clinical presentation.
Time Frame: 6 months after TBI
Measure: Mean (Standard Error); unit: weeks
Arm/Group | Placebo | Sertraline
Number analyzed (Participants) | 46 | 48
weeks | 21.4264 (0.9982) | 15.7833 (0.2091)
Statistical Analysis 1: Comparison: Placebo vs Sertraline; Test type: Superiority or Other; p < 0.05, Log Rank; Hazard Ratio (HR) = 3.6, 95% CI 2-sided [1.1 to 16.2]

2. Secondary Outcome: Total Community Integration Questionnaire Scores
Description: The Community Integration Questionnaire (CIQ) is intended as a brief, reliable measure of an individual's level of integration into the home and community following traumatic brain injury. Total CIQ scores were used as the outcome measure. Range: 0 to 25. Higher scores indicate higher levels of integration into the home and community following TBI.
Time Frame: 6 months after TBI
Population: Out of the 80 participants who completed the trial, only 68 completed CIQ at this evaluation time.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Sertraline
Number analyzed (Participants) | 30 | 38
units on a scale | 16.77 (3.69) | 17.67 (4.37)

3. Secondary Outcome: Iowa Gambling Task Score
Description: The Iowa Gambling Task (IGT) evaluates decision making ability. During IGT subjects have to choose between decks of cards which yield high immediate gain but larger future loss (i.e., long term loss), and decks which yield lower immediate gain but a smaller future loss (i.e., a long term gain). The task consists of four decks of cards: A, B, C, and D. The goal in the task is to maximize profit. Subjects are required to make a series of card selections. The decks A and B are long term loss decks and the decks C and D are long term gain decks. The IGT Score reported is the combination of the raw score for each deck combined in the following way: (C+D) - (A+B). The range for this score is: -100 to 100. Higher values of this score indicate better decision making ability.
Time Frame: 6 months after TBI
Population: Out of the 80 participants who completed the trial, only 64 completed IGT at this evaluation time.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Sertraline
Number analyzed (Participants) | 33 | 31
units on a scale | 16.67 (29) | -0.77 (28)

4. Secondary Outcome: Memory Function Composite
Description: This outcome measures memory function and is a composite of five standardized scores: Brief Visuospatial Memory Test - Revised, Delayed Recall and California Verbal Learning Test, Short Delay Free Recall Number Correct and Discriminability, and Long Delay Free Recall Number Correct and Discriminability. Standardized scores (i.e., z-scores) for each test of this composite were obtained by subtracting the mean raw score of all participants to the raw score of each participant and dividing the result by the standard deviation of the raw scores of all participants. The composite score was obtained by averaging the z-scores of the four memory tests mentioned previously. Range: -3 to 3. Higher scores represent better memory function.
Time Frame: 6 months following traumatic brain injury
Population: Out of the 80 participants who completed the trial, only 61 completed all the tests necessary to calculate the composite score at this evaluation time.
Measure: Mean (Standard Deviation); unit: z-scores
Arm/Group | Placebo | Sertraline
Number analyzed (Participants) | 29 | 32
z-scores | -0.08 (0.75) | 0.07 (0.88)

5. Secondary Outcome: Social Functioning Examination Total Score
Description: The Social Functioning Examination (SFE) is a semi-structured interview that measures social functioning in areas such as interpersonal relationships, work adjustment, use of community resources and satisfaction with living environment. Range: 0 to 1. Higher scores denote lower levels of social functioning.
Time Frame: 6 months after TBI
Population: Out of the 80 participants who completed the trial, only 63 completed SFE at this evaluation time.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Sertraline
Number analyzed (Participants) | 29 | 34
units on a scale | 0.04 (0.04) | 0.04 (0.06)

6. Secondary Outcome: Neuroimaging Variables (i.e., Fractional Anisotropy [FA] of Frontal White Matter Such as the Cingulate Gyrus)
Description: FA is a measured obtained from Diffusion Tensor Imaging, an image modality of Magnetic Resonance Imaging (MRI). FA is a unitless index. Range: 0 to 1. FA describes the degree of anisotropy of a diffusion process. A value of zero means that diffusion is unrestricted or equally restricted in all directions. A value of one means that diffusion occurs only along one axis and is fully restricted along all other directions. In the context of this study, FA measures the integrity of the cingulate gyrus white matter. Higher FA values reflect higher integrity of the cingulate gyrus white matter tract. Average FA values for the right and left cingulate gyri were summed.
  One aim of this project was to identify predictors of the occurrence of mood disturbances during the first 6 months following TBI. The hypothesis for this aim was that patients who develop a mood or anxiety disorder six months after TBI present at baseline with lower FA of the cingulate gyrus than those who do not.
Time Frame: Baseline
Population: Of the 94 participants randomized, only 61 participants had an MRI and were included in the analysis of this study aim.
Measure: Mean (Standard Deviation); unit: unitless index
Arm/Group | Patients Who Developped a Mood or Anxiety Disorder | Patients Who Did Not Developped a Mood or Anxiety Disorder
Number analyzed (Participants) | 8 | 53
unitless index | 0.91 (0.06) | 0.94 (0.07)

ADVERSE EVENTS:
Arm/Group | Placebo | Sertraline
Serious Adverse Events (participants affected / at risk) | 1/46 | 1/48
Other Adverse Events (participants affected / at risk) | 31/46 | 35/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=46) | Sertraline (N=48)
Hip fracture (Musculoskeletal and connective tissue disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=46) | Sertraline (N=48)
Diarrhea (General disorders) | 7 | 15
Dizziness (General disorders) | 9 | 12
Dry mouth (General disorders) | 2 | 12
Fatigue (General disorders) | 1 | 3
Insomnia (General disorders) | 6 | 3
Lightheadedness (General disorders) | 7 | 8
Nausea (General disorders) | 3 | 3
Sweating (General disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No